CLINICAL TRIAL: NCT02210338
Title: A Comparison of the C-mac and Bonfils Intubation Fibrescope for Tracheal Intubation in Patients With a Simulated Difficult Airway
Brief Title: A Comparison of the C-mac and Bonfils Intubation Fibrescope
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: sghan-cb01
Record Dates: First submitted 2014-08-05; First posted 2014-08-06 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Intubation; Airway

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Karl Storz C-MAC (Experimental): Intubation of patient using the Karl Storz C-MAC video laryngoscope
  Interventions: Device: Karl Storz C-MAC
- Bonfils Intubation Fibrescope (Experimental): Intubation of patient using Bonfils Intubation Fibrescope
  Interventions: Device: Bonfils Intubation Fibrescope

INTERVENTIONS:
Device: Karl Storz C-MAC
  Arms: Karl Storz C-MAC
Device: Bonfils Intubation Fibrescope
  Arms: Bonfils Intubation Fibrescope

SUMMARY:
The study aims to determine the better device to facilitate intubation in patients with a limited neck movement and small mouth opening. This may help anesthesiology as well as emergency medicine practitioners and departments to decide when choosing between these two conceptually similar device. The hypothesis to be tested is that the C-MAC® is more superior when compared to the Bonfils Intubation Fibrescope in success of intubation, time to intubation and complication rate in patients with a fixed cervical collar.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective surgery under general anaesthesia who require endotracheal intubation

Exclusion Criteria:

* Patients with history of previous difficult endotracheal intubation
* Patients with two or more predictors of difficult mask ventilation or difficult intubation or the combination of both
* Patients with ASA (American Society of Anesthesiologists) grading of III and above are excluded from the study, as well as patients with 2 or more predictors for difficult mask ventilation or difficult intubation or the combination of both.
* Patients needing a rapid sequence induction for rapid securement of the airway
* Pregnant women
* Patients below the age of 21 years old
* Patients unfit to give consent

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-12 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Success of intubation on first attempt | up to 10min - from time of induction to appearance of end tidal carbon dioxide on capnograph after first attempt at intubation
  A rigid cervical collar will to each patient to stimulate a difficult airway and standard induction of general anaesthesia will be carried out. Adequate muscle relaxation will be confirmed by the use of a standard neuromuscular Train-of-Four monitor, showing no twitch. Intubation will then proceed with the assigned airway device. A successful outcome at intubation will involve being able to pass an appropriately sized endotracheal tube pass the vocal cords into the trachea on the first try, as evidenced by the presence of end tidal carbon dioxide on a capnograph.

SECONDARY OUTCOMES:
Time taken to successful intubation | up to 10min - from time of induction to appearance of end tidal carbon dioxide on capnograph after successful intubation
  A rigid cervical collar will to each patient to stimulate a difficult airway and standard induction of general anaesthesia will be carried out. Adequate muscle relaxation will be confirmed by the use of a standard neuromuscular Train-of-Four monitor, showing no twitch. Time to successful intubation will then be measured from the first handling of the airway device, until successful intubation with an endotracheal tube is confirmed by the presence of end tidal carbon dioxide on a capnograph trace.

CONTACTS AND LOCATIONS:
Overall Officials: Theodore GL Wong, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore, Singapore

REFERENCES:
- [Background] Abdullah HR, Li-Ming T, Marriott A, Wong TG. A comparison between the Bonfils Intubation Fiberscope and McCoy laryngoscope for tracheal intubation in patients with a simulated difficult airway. Anesth Analg. 2013 Nov;117(5):1217-20. doi: 10.1213/ANE.0b013e3182a46fa9. PMID 24029854